CLINICAL TRIAL: NCT00002300
Title: Phase II-III Randomized Double-Blind Study Comparing Megestrol Acetate at 100, 400, and 800 mg/Day, and Placebo in AIDS Patients With Anorexia and Cachexia
Brief Title: A Study of Different Doses of Megestrol Acetate in Patients With AIDS Who Have Anorexia and Malnutrition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 025A; MEG8807
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-10

CONDITIONS: Anorexia; Cachexia; HIV Infections
Keywords: T-Lymphocytes; Megestrol; Dose-Response Relationship, Drug; Acquired Immunodeficiency Syndrome; Anorexia; Cachexia
MeSH Terms: conditions — Anorexia; Cachexia; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Megestrol Acetate

INTERVENTIONS:
Drug: Megestrol acetate

SUMMARY:
To compare the effects of megestrol acetate and placebo on body weight, anorexia, cachexia, calorie intake, and nutritional parameters of patients with a confirmed diagnosis of AIDS. To characterize dose response in relation to weight gain. To determine whether megestrol acetate relative to placebo improves the perception of well-being among AIDS patients with cachexia. To evaluate megestrol acetate's effect on immune function via skin test reactivity, T4/T8 ratio, and total lymphocytes.

ELIGIBILITY:
Inclusion Criteria

Patient must have:

* Confirmed diagnosis of AIDS (CDC definition).
* Documented weight loss or anorexia.
* Life expectancy = or > 20 weeks.
* The perception that the weight loss is a detriment to their well-being.
* Ability to provide informed consent, read and write English.

Prior Medication:

Allowed:

* Ganciclovir.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Dementia or evidence of mental incompetence which would preclude compliance with the protocol.
* Diarrhea defined as 5 or more watery stools per day for at least 7 days.
* Active uncontrolled systemic infections at the start of treatment.
* (Patients may not be entered for at least 2 weeks after acute infection.) Clinical or radiologic evidence of ascites or pleural effusions.

Concurrent Medication:

Excluded:

* Therapy designed to treat the underlying HIV infection or which may have a major impact on appetite and/or weight gain.
* Patients who have been started on zidovudine (AZT) within eight weeks. (Patients may have been previously treated with AZT and failed or may currently be receiving AZT for at least 8 weeks.)

Patients with the following are excluded:

* Obstruction to food intake or impaired digestive/absorptive functions.
* Contraindications to high-dose megestrol acetate (poorly controlled hypertension or heart failure or deep vein thrombosis).
* Inability to consent or be available for close follow-up.
* Active systemic infections at the start of treatment.
* Patients may not be started on any therapy designed to treat the underlying HIV infection or which may have a major impact on appetite and/or weight gain.
* Clinical or radiologic evidence of ascites or pleural effusions.
* Patients may not be started on any therapy designed to treat the underlying HIV infection or which may have a major impact on appetite and/or weight gain.
* Patients who have been hospitalized or have suffered an exacerbation of their illness associated with weight loss within the past 2 weeks are excluded.
* Menstruating female patients are excluded.

Prior Medication:

Excluded:

* Corticosteroids.
* Anabolic steroids.
* Marijuana.
* Megestrol acetate.
* Patients who have been started on zidovudine (AZT) within 8 weeks. (Patients may have been previously treated with AZT and failed or may currently be receiving AZT for at least 8 weeks.) History of substance abuse and questionable current and future abstinence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Birmingham Veterans Administration Med Ctr / Univ of Alabama, Birmingham, Alabama
  - Dr NS Tchekmedyian, Long Beach, California
  - Dr Stephen J Gabin Jr, Los Angeles, California
  - Eisenhower Med Ctr, Rancho Mirage, California
  - Denver Public Health Dept, Denver, Colorado
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Veterans Administration Med Ctr, Washington D.C., District of Columbia
  - Miami Veterans Administration Med Ctr, Miami, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - Albany Med College / AIDS Treatment Ctr, Albany, New York
  - Community Research Initiative on AIDS, New York, New York
  - Saint Vincent's Hosp and Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Audie L Murphy Veterans Administration Hosp, San Antonio, Texas

REFERENCES:
- [Background] Strang P. The effect of megestrol acetate on anorexia, weight loss and cachexia in cancer and AIDS patients (review). Anticancer Res. 1997 Jan-Feb;17(1B):657-62. PMID 9066597